CLINICAL TRIAL: NCT04263298
Title: A Randomized, Multi-center, Open-label, Phase III Trial of Fulvestrant Versus Capecitabine as Maintenance Therapy After First-line Chemotherapy in Patients With Hormone Receptor Positive, Human Epidermal Growth Factor Receptor-2 Negative Metastatic Breast Cancer (FAMILY)
Brief Title: Fulvestrant Versus Capecitabine as Maintenance Therapy After First-line Chemotherapy in Patients With HR+/HER2- Metastatic Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Herui Yao (Other)
Responsible Party: Sponsor-Investigator, Herui Yao, Principal Investigator, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Organization: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYS-C-201801-5010
Record Dates: First submitted 2020-02-04; First posted 2020-02-10 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fulvestrant Group (Experimental): Fulvestrant 500mg Days 0, 14, 28, then every 28 days
  Interventions: Drug: Fulvestrant
- Capecitabine Group (Active Comparator): Capecitabine 2000mg/m2 twice daily x 14 days followed by 7 days off
  Interventions: Drug: Capecitabine Oral Product

INTERVENTIONS:
Drug: Fulvestrant — Fulvestrant 500mg Days 0, 14, 28, then every 28 days
  Other Names: Experimental group
  Arms: Fulvestrant Group
Drug: Capecitabine Oral Product — Capecitabine 2000mg/m2 twice daily x 14 days followed by 7 days off
  Other Names: Active Comparator control group
  Arms: Capecitabine Group

SUMMARY:
This phase III trial aims to compare the efficacy and safety of fulvestrant or capecitabine as maintenance therapy after first-line chemotherapy in hormone receptor-positive, human epidermal growth factor receptor-2 negative metastatic breast cancer.

DETAILED DESCRIPTION:
Metastatic breast cancer (MBC) is incurable. Although first-line endocrine therapy is preferred to hormone receptor positive (HR+), human epidermal growth factor receptor-2 negative (HER2-) MBC, chemotherapy may be reserved as the initial treatment for patients with rapid clinical progression, life-threatening visceral metastases, and need for rapidly symptom control. Either prolonged chemotherapy or endocrine therapy may be used as maintenance after disease control. However, which maintenance strategy is superior in terms of delaying disease progression as well as maintaining quality of life (QOL) remains uncertain. This phase III trial aims to compare the efficacy and safety of fulvestrant or capecitabine as maintenance therapy after first-line chemotherapy in HR+/HER2- MBC.

ELIGIBILITY:
Inclusion Criteria:

* Adult female patients with advanced breast cancer diagnosed by pathology (aged 18-75, including 18 and 75 years old), not suitable for surgical resection or radiation therapy for the purpose of cure;
* Pathological examination confirmed ER and / or PR positive, HER-2 negative (Positive ER expression: immunohistochemistry >1% tumor cell staining; Positive PR expression: immunohistochemistry >1% tumor cell staining; HER-2 negative: immunohistochemistry is 0,1+, or FISH/CISH negative when immunohistochemistry is 2+);
* Patients with advanced breast cancer who have no disease progression after a 4-8-course first-line chemotherapy regimen (the effect is evaluated as complete response/ partial response/ stable disease). Capecitabine monotherapy as first-line chemotherapy is allowed and the courses of treatment should be limited to 6.
* WHO physical status 0-1 points, estimated lifetime at least 3 months;
* Imaging examinations within 3 weeks before enrollment were required for assessing tumor lesions before maintenance treatment (Examination results from local Tertiary A hospital are available);
* Previous treatment-related toxicity should be relieved to ≤ Grade 1 according to NCI CTCAE (version 4.03) before randomization (Except for hair loss and other toxicities that are not at risk to the patient's safety based on the investigator's judgment);
* The routine blood test was normal within 1 week before enrollment: WBC ≥3.0×10^9／L, b. ANC ≥1.5×10^9／L, c. PLT ≥100×10^9／L;
* The liver and kidney function test was normal within 1 week before enrollment (Take the normal value of the laboratory of each research center as the standard): a. TBIL≤1.5× Upper Limit of Normal (ULN)b. ALT/AST≤2.5×ULN（Liver metastasis patients ≤5xULN） c. Serum Cr ≤1.5×ULN, or Ccr ≥60 ml/min;
* Informed consent form signed before enrollment.

Exclusion Criteria:

Cannot be grouped if any of the following is true:

* Newly developed central nervous system metastasis or symptom control of central nervous system is less than 4 weeks. (Patients with asymptomatic brian metastases which was stable more than 4 weeks by imaging assessment and do not need corticosteroid therapy are allowed to enrollment)
* Diagnosis of any other malignant tumor within 3 years before randomization, except for adequately treated basal cells or squamous cell skin cancer or cervical cancer in situ;
* Endocrine therapy for advanced disease;
* Pregnant or breast-feeding patients;
* Patients with accompanying disease or situation that may interfere with the study, or any serious medical problems that may affect the safety of the subject (for example, uncontrolled heart disease or high blood pressure, active or uncontrolled infection, active hepatitis B virus infection);
* Patients who were unable to tolerate capecitabine toxicity were first identified in first-line treatment;
* Patients with recurrent metastatic disease within 2 years of adjuvant endocrine therapy (including 2 years);

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2030-05-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Estimated 18 months
  From enrollment to progression or death (for any reason)

SECONDARY OUTCOMES:
Overall Survival (OS) | Estimated 60 months
  From enrollment to death (for any reason)
Objective Response Rate (ORR) | Estimated 18 months
  Ratio of CR and PR in all subjects
Clinical Benefit Rate (CBR) | Estimated 18 months
  Ratio of CR,PR and SD greater than or equal to 24 weeks in all subjects
Quality Of Life (QOL) | Estimated up to 60 months
  All patients need to fill in the Functional Assessment of Cancer Therapy-Breast (FACT-B), a 44-item self-report instrument designed to measure multidimensional quality of life (QL) in patients with breast cancer.
Adverse Events and Serious Adverse Events | From informed consent through 28 days following treatment completion
  Safety

CONTACTS AND LOCATIONS:
Overall Officials: Herui Yao, PhD, Study Chair — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University; Shusen Wang, PhD, Principal Investigator — Sun Yat-sen University; Kun Wang, PhD, Principal Investigator — Guangdong Provincial People's Hospital; Peijian Peng, PhD, Principal Investigator — Fifth Subsidiary Sun Yat-sen University Hospital; Li Ling, PhD, Principal Investigator — Public Health Institute of Sun Yat-sen University; Yongkui Lu, MD, Principal Investigator — Affiliated Cancer Hospital of Guangxi Medical University; Quchang Ouyang, PhD, Principal Investigator — Hunan Cancer Hospital; Ying Lin, phD, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University; Ying Zhang, MD, Principal Investigator — Affiliated Hospital of Guangdong Medical University; Mei Huang, MD, Principal Investigator — The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine; Zhiyong Wu, MD, Principal Investigator — Shantou Central Hospitalv; Cai'wen Du, PhD, Principal Investigator — Chinese Academy of Medical Sciences
Locations (13):
- China (13):
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Public Health Institute of Sun Yat-sen University, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Shantou Central Hospital, Shantou, Guangdong
  - Cancer Hospital, Chinese Academy of Medical Sciences, Shenzhen Center, Shenzhen, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Affiliated Hospital of Guangdong Medical University, Zhangjiang, Guangdong
  - Fifth Subsidiary Sun Yat-sen University Hospital, Zhuhai, Guangdong
  - Affiliated Cancer Hospital of Guangxi Medical University, Nanning, Guangxi
  - Hunan Cancer Hospital, Changsha, Hunan

IPD SHARING:
Plan to Share IPD: No